CLINICAL TRIAL: NCT04041752
Title: Satietogenic Effect of Liquid Versus Solid Meals in Healthy Adults
Brief Title: Meal Texture and Satiety
Acronym: FEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Appetite Control and Energy Balance Research Group, UNiversity of Leeds, Leeds, UK (Unknown); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2018 BOIRIE 2; 2019-A00033-54 (Other: 2019-A00033-54)
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Healthy Normal Weight
Keywords: Meal texture; Appetite; Energy compensation; Food reward

STUDY DESIGN:
Intervention Model Description: All participants complete the same conditions
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal weight (Experimental): 30 healthy normal weight adults will be involved and will realize the three conditions
  Interventions: Behavioral: SOLID; Behavioral: LIQUID_P; Behavioral: LIQUID_L

INTERVENTIONS:
Behavioral: SOLID — condition with a classical meal served using solid food items
Behavioral: LIQUID_P — condition with a liquid meal served using a powder solution
Behavioral: LIQUID_L — condition with a pre-prepared meal served using a liquid solution.

SUMMARY:
The aim of the present study is to compare the nutritional compensation between iso-caloric meals of various textures (liquid vs solid) in health young adults.

DETAILED DESCRIPTION:
The present study will compare the potential energy intake compensations, appetite feelings response, food reward variations and satiating responses after the ingestion of three different lunch meals: i) one classical cooked meal; ii) one iso-energetic meal consumed using a pre-prepared liquid meal; iii) one iso-energetic meal consumed using a prepared liquid meal. This will be the first study to assess all these nutritional factors after such meals.

ELIGIBILITY:
Inclusion Criteria:

* being aged 18 to 25 years old
* Being normal weight with a BMI between 20 and 25 kg/m²
* Being registered with a social security number

Exclusion Criteria:

* Eating disorders
* Specific food allergies or habits
* being under diet

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Spontaneous Energy intake measured | day 1 , day 8, day 15
  spontaneous food intake will be measured ad libitum for the 12 hours that will follow the laboratory sessions (between 02:00pm to 11:59 pm). The participants will be offered a food bag composed of items they like and proposed ad libiutm and will be asked to only conume food from this bag for the rest of the day. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using Bilnuts software.

SECONDARY OUTCOMES:
Hunger feelings | day 1 , day 8, day 15
  hunger area under the curve will be assessed using visual analogue scale through a the day
Food reward | day 1 , day 8, day 15
  The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ)

CONTACTS AND LOCATIONS:
Overall Officials: yves Boirie, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France